CLINICAL TRIAL: NCT00988078
Title: Effect of Metformin Therapy on Insulin Resistance and Melatonin in Adolescents With Polycystic Ovary Syndrome.
Brief Title: Effects of Metformin and Oral Hormonal Contraceptive in Adolescents With Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Margareth Chiharu Iwata, post graduation, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 2102/08
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2009-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: metformin; Hyperandrogenism; Metabolic Syndrome X; adolescents; melatonin; Polycystic Ovary Syndrome; Insulin Resistance; Menstrual Cycle
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Metabolic Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin 500mg three times a day for six months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): 1 capsule three times a day for six months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Capsule (without biologic action) administered three times a day for six months
  Arms: Placebo
Drug: Metformin — Metformin 500mg three times a day for six months
  Arms: Metformin

SUMMARY:
The polycystic ovary syndrome is the most common endocrinopathy in reproductive age women. The pathophysiology of this syndrome remains unclear, but there are evidences that a decreased in insulin sensitivity may be related in this syndrome. There are studies that showed the action of factors on the sensitivity of the insulin receptor, such as melatonin. It is a hormone produced by the pineal gland, whose role is still uncertain in human reproduction, although many studies have found that it may relate sex hormone effect. Many patients with polycystic ovary syndrome (PCOS) may have hyperinsulinemia, and that pinealectomized rats determined hypoglycemia and hyperinsulinemia, with reduced release of insulin in response to glucose. Therefore, it is supposed that blood levels of melatonin might correlate with the blood insulin concentration in patients with the syndrome. Moreover, the insulin sensitizing agents have been used in the treatment of patients with insulin resistance and PCOS, based on its main pathophysiological substrate which is the hyperinsulinemia. In fact, the metformin is the most used in the literature. However, there are few studies on the use of metformin in adolescents. The evidences of this drugs in this group of patients have showed good therapeutic response with few side effects. The objective of the study is to evaluate the effects of metformin on insulin resistance and levels of melatonin in adolescents with PCOS. It will be performed a prospective, randomized, double-blind and placebo-controlled study with 90 adolescents with PCOS. It will be evaluated clinical and laboratory parameters (TSH, free T4, prolactin, FSH, LH, estradiol, total testosterone, androstenedione, DHEA-s, 17-OH progesterone, SHBG, free androgen index, index of HOMA-IR and QUICKI from fasting glucose and insulin, total cholesterol and fractions, triglycerides, creatinine, AST and ALT and creatinkinase, fibrinogen and PAI-1, and melatonin for 6 months of treatment.

DETAILED DESCRIPTION:
Design: 90 patients will be selected to a prospective, randomized and double-blinded study. They will be assigned to two groups: A) 45 patients, treated with OC (oral contraceptive) and metformin 1500mg/ day. B) 45 patients, treated with OC and placebo. The length of treatment was six months.

Inclusion criteria: patients until 19 years-old, at least 2 years after menarche, with Polycystic Ovary Syndrome based on Rotterdan criterion. Exclusion criteria: patients with Diabetes Mellitus, hypertension, hyperprolactinemia, adrenal enzymatic deficiency, Cushing syndrome, thyroidopathy, renal or hepatic disfunction, use of OC or insulin-sensitising drugs in the last 90 days before, pregnancy, androgen tumors, hormonal-sensitive tumors in the past, contra-indication to the medications used in the study.

Clinical parameters included are weight and height (for BMI), waist to hip ratio, habits like smoking or drinking, drug addiction, blood pressure measurement, hirsutism and acne.

Laboratorial parameters included are TSH, free T4, prolactin, FSH, LH, estradiol, total testosterone, androstenedione, s-DHEA, 17-OH progesterone, SHBG, free androgen index, fasting glucose and insulin, total cholesterol and fractions, triglycerides, creatinin, TGO, TGP, CK, PAI-1, fibrinogen, melatonin.

Patients will be evaluated using these parameters in the beginning, 1, 3 and 6 months after use of the drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients until 19 years-old, at least 2 years after menarche
* Patients with Polycystic Ovary Syndrome based on Rotterdan criteries

Exclusion Criteria:

* Patients with Diabetes Mellitus, hypertension, hyperprolactinemia, adrenal enzymatic deficiency, Cushing syndrome, thyroidopathy, renal or hepatic disfunction
* Use of OC or insulin-sensitising drugs in the last 90 days before
* Pregnancy
* Androgen tumors, hormonal-sensitive tumors in the past
* Contra-indication to the medications used in the study

Ages: 11 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
serum melatonin | 0 and 6 months

SECONDARY OUTCOMES:
hormonal and metabolic measurements, clinical assessment | 0, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Soares Junior, Study Director — Federal University os Sao Paulo; Alexandre Rossi, Study Chair — Federal University os Sao Paulo; Eduardo Leme Alves da Motta, Study Director — Federal University os Sao Paulo; Margareth Chiharu Iwata, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil